CLINICAL TRIAL: NCT03085433
Title: Sperm Selection by Microfluidic Separation Improves Embryo Quality
Acronym: SPERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-21273
Record Dates: First submitted 2017-03-19; First posted 2017-03-21 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Sperm DNA Fragmentation; Embryo Quality; Fertility Disorders; Infertility; Infertility, Male; Infertility Unexplained
MeSH Terms: conditions — Infertility; Infertility, Male | interventions — Fertilization in Vitro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Microfluidic sperm sorting (Experimental): Couples undergoing in vitro fertilization randomized to microfluidic sperm sorting will have raw semen sorted by the microfluidics chip prior to fertilization with IVF/ICSI.
  Interventions: Device: Microfluidic Sperm Sorting; Procedure: in vitro fertilization
- Conventional sperm preparation (Active Comparator): Couples undergoing in vitro fertilization randomized to conventional methods for sperm processing will undergo separation of semen by density gradient centrifugation prior to IVF/ICSI.
  Interventions: Procedure: in vitro fertilization

INTERVENTIONS:
Device: Microfluidic Sperm Sorting — Microfluidic technology isolates healthy sperm by laminar flow, creating gradients through channels. The microfluidic chip we plan to study in our randomized clinical trial utilizes space-constrained microfluidic sorting to select highly motile and morphologically normal sperm in a flow and chemical-free design. Unlike the standard of density gradient centrifugation, no manipulation of sperm is required in this process. Raw semen is introduced into the inflow and only motile and morphologically normal sperm are able to swim through the chip to the outflow where it is collected for use.
  Other Names: FERTILE device
  Arms: Microfluidic sperm sorting
Procedure: in vitro fertilization — ivf/icsi

SUMMARY:
This is a randomized controlled trial of couples with a history of poor embryo quality undergoing a repeat in vitro fertilization (IVF) cycle for unexplained infertility. Couples will be randomized to sperm selection by the clinical standard of centrifugation and density-gradient processing compared to the microfluidic sperm sorting chip.

DETAILED DESCRIPTION:
More than 70 million couples worldwide are infertile and up to 40 million are actively seeking infertility care. In the year 2013, a total of 160,521 assisted reproductive technology (ART) procedures were performed in the United States. Isolation of motile and morphologically normal sperm is an integral part of assisted reproduction. Traditional sperm processing for assisted reproduction involves centrifugation and "swim up" techniques that employ a density gradient to isolate motile sperm. This technique involves several steps of centrifugation (200-1800g) with colloidal silica particles. In this process, sperm and other material form distinct bands. It is thought that this procedure allows for elimination of abnormal/immotile sperm as well as debris, thereby isolating motile human sperm. Nevertheless, the centrifugation process has been shown to induce DNA damage and produce reactive oxygen species, thereby potentially compromising sperm quality and subsequent laboratory outcomes such as fertilization rate and embryo quality. Increased sperm DNA damage has been associated with poor outcomes in assisted reproduction, including lower fertilization rates, impaired embryo progression, and decreased pregnancy rates. The details of the density gradient centrifugation process are not regulated by the FDA.

In contrast, microfluidic-based sperm sorting has the capability of selectively isolating highly motile, morphologically normal sperm with high DNA integrity from an unprocessed semen sample. Microfluidic technology isolates healthy sperm by laminar flow, creating gradients through channels. The microfluidic chip we plan to study in our randomized clinical trial utilizes space-constrained microfluidic sorting to select highly motile and morphologically normal sperm in a flow and chemical-free design. Unlike the standard of density gradient centrifugation, no manipulation of sperm is required in this process. Raw semen is introduced into the inflow and only motile and morphologically normal sperm are able to swim through the chip to the outflow where it is collected for use.

In semen samples from healthy male volunteers split into standard processing via centrifugation and swim-up procedure compared with microfluidic sperm sorting, a significantly higher percent motility and lower rate of sperm DNA fragmentation was detected with microfluidic sperm sampling. The microfluidic sperm sorting technique has thus proven to be an efficient and reliable means of sperm preparation compared with the centrifugation and swim-up procedure. While this microfluidic chip has been used clinically in Mexico, Turkey, South Africa, Italy, Greece, and Switzerland resulting in over 5,000 live births, its use in clinical practice has not been rigorously studied. We aim to compare traditional preparation and microfluidic sperm sorting on assisted reproductive technology outcomes including oocyte fertilization and embryo quality in subjects with a history of poor embryo quality electing to undergo a repeat in vitro fertilization cycle for infertility.

ELIGIBILITY:
Inclusion Criteria:

* The target population includes couples planning in vitro fertilization (IVF) with intracytoplasmic sperm injection (ICSI).
* Subjects with and without a history of prior IVF cycles will be included.
* All eligible couples where both partners are >=18 years of age will be asked to join the study.

Exclusion Criteria:

* Male partner with severe oligoasthenospermia (concentration < 5 x 10^6 spermatozoa/mL; motility< 10%)
* Female partner with anovulation (PCOS, FHA)
* Female partner age >41
* Female partner AFC< 7
* Female partner with obstructed fallopian tubes (assessed in all patients prior to IVF)
* Use of oocyte donor
* Either Partner:

  * Cancer diagnosis in either partner
  * Any significant disease or psychiatric disorder that would interfere with consenting process
* Treatment History:

  o History of >1 prior cycle cancellation due to poor response
* Treatment Plan:

  * Embryo co-culture
  * Use of adjunctive non-gonadotropin medications to improve embryo quality: growth hormone, sildenafil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Rosen, M.D, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quinn MM, Ribeiro S, Juarez-Hernandez F, Simbulan RK, Jalalian L, Cedars MI, Rosen MP. Microfluidic preparation of spermatozoa for ICSI produces similar embryo quality to density-gradient centrifugation: a pragmatic, randomized controlled trial. Hum Reprod. 2022 Jun 30;37(7):1406-1413. doi: 10.1093/humrep/deac099. PMID 35522187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between June 2017 and September 2021. All patients were screened at the time of consultation for eligibility. During this time frame, 1190 patients were eligible to participate and 393 consented to participation.
Pre-assignment Details: 7 consented participants either voluntarily withdrew from the study or their fertility treatment cycles were cancelled prior to randomization. Ultimately 386 participants were randomized to intervention assignments.
Period: Overall Study
Arm/Group | Microfluidic Sperm Sorting | Conventional Sperm Preparation
Started | 192 | 194
Completed | 157 (35 did not participate in assigned arm due to patient request to widthdraw post randomization or physician deemed clinical necessity to alter plan to optimize clinical success and participant was no longer eligible per study protocol and design.) | 140 (54 did not participate in assigned arm due to patient request to widthdraw post randomization or physician deemed clinical necessity to alter plan to optimize clinical success and participant was no longer eligible per study protocol and design.)
Not Completed | 35 | 54
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Physician Decision | 33 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Microfluidic Sperm Sorting | Conventional Sperm Preparation | Total
Number analyzed (Participants) | 157 | 140 | 297
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 157 | 140 | 297
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (4.6) | 38.4 (5.7) | 38.4 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 157 | 140 | 297
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 157 | 140 | 297
Region of Enrollment [Number; unit: participants]
  United States | 157 | 140 | 297

OUTCOME MEASURES:

1. Primary Outcome: Day 3 High Quality Embryo Percentage
Description: The primary outcome for intent to treat analysis. Day 3 high quality embryo percentage rate will be defined as the percentage of all viable 2PN embryos on day 3 with at least 6 cells and fragmentation/symmetry scores of 1-2. Scale: 1-6 for either fragmentation or symmetry. Lower scores are better. Calculated as ( the number of high-qualify-grade embryos yielded by a participant / the number of all viable 2PN embryos yielded by the participant x 100)
Time Frame: 3 days following fertilization
Population: Embryo grade 6c or greater, <10% fragmentation, symmetry: even/slightly uneven will be considered "high quality".
Measure: Mean (Standard Deviation); unit: percentage of high quality embryos
Arm/Group | Microfluidic Sperm Sorting | Conventional Sperm Preparation
Number analyzed (Participants) | 157 | 140
percentage of high quality embryos | 68 (30.3) | 66 (25.8)

2. Secondary Outcome: Egg Fertilization Rate
Description: Number of eggs successfully fertilized (2PN embryo count) per number of mature eggs (MII egg count) retrieved per participant. 2PN grade indicates a successfully fertilized embryo. MII grade indicates a metaphase II stage egg which is mature enough to undergo fertilization. (The percentage is calculated for each participant as the number of 2PN embryos obtained / the number of MII eggs obtained x100). The resulting percentages were then averaged to determine the average fertilization rate for participants in each study arm.
Time Frame: 1 day following fertilization
Measure: Mean (Standard Deviation); unit: percentage of eggs that fertilized
Arm/Group | Microfluidic Sperm Sorting | Conventional Sperm Preparation
Number analyzed (Participants) | 157 | 140
percentage of eggs that fertilized | 75.2 (17.8) | 79.4 (19.4)

3. Secondary Outcome: Pregnancy Rate
Description: Pregnancy rate will be defined as achieving a clinical pregnancy ( an ultrasound demonstrating gestational sac with yolk sac) per embryo transfer procedure attempt.
Time Frame: 14 days following embryo transfer
Measure: Count of Participants; unit: Participants
Arm/Group | Microfluidic Sperm Sorting | Conventional Sperm Preparation
Number analyzed (Participants) | 157 | 140
Participants | 82 | 78

ADVERSE EVENTS:
Time Frame: Adverse event data for participants was collected over a period of 2weeks.
Arm/Group | Microfluidic Sperm Sorting | Conventional Sperm Preparation
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/140
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/140
Other Adverse Events (participants affected / at risk) | 0/157 | 0/140

LIMITATIONS AND CAVEATS:
The population studied was inclusive and did not attempt to isolate male factor infertility cases or patients with a history of elevated sperm DNA fragmentation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT03085433/Prot_SAP_002.pdf
  • Informed Consent Form (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT03085433/ICF_003.pdf